CLINICAL TRIAL: NCT04542161
Title: Mechanistic Assessment of N-Acetylcysteine as an Antioxidant Therapy for Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) Through Dose Response and Treatment Target Engagement
Brief Title: Assessment of N-Acetylcysteine as Therapy for Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Acronym: NAC ME/CFS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20-01021280; R01NS116887 (NIH)
Record Dates: First submitted 2020-08-28; First posted 2020-09-09 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NAC 900mg/day (Active Comparator): Subjects who pass screening may be randomly assigned to this arm where they will self administer NAC 900mg/day caplets for a four week period
  Interventions: Drug: NAC 900mg/day
- NAC 3600mg/day (Active Comparator): Subjects who pass screening may be randomly assigned to this arm where they will self administer NAC 3600mg/day caplets for a four week period
  Interventions: Drug: NAC 3600mg/day
- NAC 0mg/day (Placebo) (Placebo Comparator): Subjects who pass screening may be randomly assigned to this arm where they will self administer NAC 0mg/day (placebo) caplets for a four week period
  Interventions: Drug: NAC 0mg/day (Placebo)

INTERVENTIONS:
Drug: NAC 900mg/day — self administer NAC 900mg/day caplets for a four week period
  Arms: NAC 900mg/day
Drug: NAC 3600mg/day — self administer NAC 3600mg/day caplets for a four week period
  Arms: NAC 3600mg/day
Drug: NAC 0mg/day (Placebo) — self administer NAC 0mg/day (placebo) caplets for a four week period
  Arms: NAC 0mg/day (Placebo)

SUMMARY:
Chronic fatigue syndrome/myalgic encephalomyelitis (ME/CFS) is an unexplained multisymptom/multisystem disorder for which there are currently no validated treatments. The present exploratory clinical trial aims to advance our understand of the mechanisms of in situ GSH synthesis control through assessment of the response of brain GSH and plasma markers of oxidative stress to different doses of NAC in comparison to placebo, as a potential treatment for ME/CFS that would provide neuroprotection against oxidative stress by restoring cortical GSH reserves. If successful, this exploratory clinical trial would address a significant public health concern by shedding new light onto the mechanisms of action of NAC in brain GSH restoration, which could open a new avenue for the development of potentially effective treatments for a disorder, ME/CFS, that currently has none.

DETAILED DESCRIPTION:
This phase two, single-site study will utilize a double-blind, placebo-controlled, randomized, pre-/post-treatment design to investigate the effect of NAC dosing on brain GSH levels and measure temporally concordant plasma levels of several established circulating markers of oxidative stress. Three study groups, of 20 subjects each (for a total of 60 who completed all components of the study), will each be administered a different dose (0 mg/day, 900mg/day, 3600mg/day) of the study intervention over a four week period; N-acetylcysteine (NAC) treatment. Subjects receiving 0 mg/day dose will be administered a placebo. Baseline visit assessments will include blood collection, survey questionnaires, MRI and MRS imaging. Subjects whose initial screening confirms low GSH level at baseline will be provided with a 4-week supplement of anonymized NAC or placebo caplets. After 4 weeks, subjects will then undergo a follow-up visit to repeat the baseline assessments.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ages 21 to 60 years (inclusive).
* Baseline GSH levels at or less than a predefined cutoff value.
* Primary diagnosis of myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS).
* Willing and capable of providing informed consent.

Exclusion Criteria:

* Significant and/or comorbid axis I (especially mood and anxiety) and axis II disorders.
* Any significant neurological illness or impairment.
* Other unstable medical conditions (asthma, hypertension, endocrine or metabolic disease, etc).
* History alcohol abuse.
* Positive urine toxicology at screening and on days of assessments.
* Positive pregnancy test at screening or on days of assessments.
* Contra-indication for clinical MRI scan (e.g., pacemaker, metallic prosthesis).
* Baseline GSH levels higher than a predefined cutoff value.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in GSH levels of treatment response: measure 1 | pre/post 4 weeks of NAC supplementation
  Levels of occipital cortex GSH, as measured in vivo with 1H MRS
Change in GSH levels of treatment response: measure 2 | pre/post 4 weeks of NAC supplementation
  Levels of striatal GSH, as measured in vivo with 1H MRS

SECONDARY OUTCOMES:
Change of levels of ventricular CSF lactate of treatment response | pre/post 4 weeks of NAC supplementation
  Levels of ventricular CSF lactate, as measured in vivo with 1H MRS
Change of regional cerebral blood flow (rCBF) of treatment response | pre/post 4 weeks of NAC supplementation
  Regional cerebral blood flow (rCBF), as measured in vivo with perfusion MRI
Change in Oxidative stress levels of treatment response: measure 1 | pre/post 4 weeks of NAC supplementation
  Level of F2-isoprostanes, a marker of oxidative stress, in plasma samples obtained
Change in Oxidative stress levels of treatment response: measure 2 | pre/post 4 weeks of NAC supplementation
  Level of 8-hydroxy-2-deoxy guanosine (8-OH-2dG), a DNA damage marker, in plasma samples obtained
Change in Oxidative stress levels of treatment response: measure 3 | pre/post 4 weeks of NAC supplementation
  Level of reduced (GSH) glutathione, an antioxidant capacity and redox state marker, in plasma obtained
Change in Oxidative stress levels of treatment response: measure 4 | pre/post 4 weeks of NAC supplementation
  Level of oxidized (GSSG) glutathione, an antioxidant capacity and redox state marker, in plasma obtained
Change in Oxidative stress levels of treatment response: measure 5 | pre/post 4 weeks of NAC supplementation
  Level of GSH peroxidase, an antioxidant enzyme activity marker, in plasma obtained
Change in Oxidative stress levels of treatment response: measure 6 | pre/post 4 weeks of NAC supplementation
  Level of protein carbonyls, a protein damage marker, in plasma obtained

CONTACTS AND LOCATIONS:
Overall Officials: Dikoma C. Shungu, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No